CLINICAL TRIAL: NCT04174924
Title: Molecular Background of Endothelial Cell Loss in Patients With Phakic Intraocular Lenses (MoBack-ECL): a Tear and Aqueous Humour Analysis Study
Brief Title: Molecular Background of Endothelial Cell Loss in Patients With Phakic Intraocular Lenses: a Tear and Aqueous Humour Analysis Study
Acronym: MoBack
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL70342.068.19
Record Dates: First submitted 2019-11-15; First posted 2019-11-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Cataract; Phakic Intraocular Lens Explantation
MeSH Terms: conditions — Cataract | interventions — Phakic Intraocular Lenses; Device Removal; Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phakic intraocular lens (pIOL) explantation: Patients with pIOLs where a combined pIOL explantation and cataract surgery is needed.
  Interventions: Procedure: Phakic intraocular lens (pIOL) explantation
- Cataract extraction: Healthy control group of patients scheduled for regular cataract surgery without comorbidities affecting an immune response.

INTERVENTIONS:
Procedure: Phakic intraocular lens (pIOL) explantation — Phakic intraocular lens (pIOL) explantation is a surgical procedure to remove the pIOL which needs to be done after cataract formation.
  Cataract extraction is a surgical procedure to remove a lens in the eye that has become cloudy over time, affecting vision in that eye.
  Other Names: Cataract extraction
  Groups: Phakic intraocular lens (pIOL) explantation

SUMMARY:
Rationale: The number of highly myopic patients is increasing. Especially in East and Southeast Asia, up to 90% of adolescents are currently myopic. Long-term treatment of high myopia can be obtained by three types of surgery: laser refractive surgery, phakic intraocular lens (pIOL) implantation, and refractive lens exchange Implantation with a pIOL is the preferred treatment for high myopes, resulting in increasing patient numbers implanted due to the increasing numbers of patients with high myopia.

Long-term results show that implantation of a pIOL induces an accelerated decrease in corneal endothelial cells (EC). Although some risk factors for increase EC loss have been identified, the underlying mechanism is currently unknown. It is hypothesized that the aqueous flow in the anterior segment of the eye (i.e. anterior chamber) is disturbed, causing an altered nutritional flow in the anterior chamber. Another hypothesis is that the pIOL causes chronic subclinical inflammation in the anterior chamber resulting in increased EC loss. Currently there is insufficient proof to confirm or reject either hypothesis. If one of these hypotheses can be confirmed, it is likely to induces significant changes in clinical practice.

Objective: The primary objective of the study is to explore the role of inflammation in the anterior chamber on endothelial cell loss in patients implanted with iris-fixated pIOLs. The secondary objective is to identify whether there is a correlation between biomarkers in aqueous humour and biomarkers in tears, both related to the accelerated progression of EC loss.

Study design: Two strategies are incorporated in the design of this study. The first part will retrospectively evaluate EC loss in patients with iris-fixated (IF) phakic intraocular lenses (pIOLs). The second part is prospective and will compare EC measurements, cytokines in aqueous humour and in tears from patients scheduled for IF-pIOLs explantation and compare them to patients with routine cataract surgery.

Study population: Patients over 18 years of age, undergoing regular cataract surgery, and patients undergoing pIOL explantation in combination with cataract surgery. A total number of 126 patients is needed, equally divided over two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Cataract in one or both eyes, or indication for pIOL explantation
* Informed and having given informed consent.

Exclusion Criteria:

* Insufficient understanding of the Dutch language to comply with study procedures
* Inability to complete follow-up or comply with study procedures
* Non-routine cataract surgery
* Cognitive or behavioral conditions that might interfere with surgery
* Patients with ocular comorbidities such as
* Women who are pregnant or nursing their child
* Immune-compromised patients (e.g., systemic corticosteroid use, leukaemia)
* Factors that increase the risk of complicated surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups will be included to compare endothelial cell loss due to inflammation in affected (i.e. iris-fixated [IF] phakic intraocular lens [pIOL] implanted) versus healthy (i.e. scheduled for regular cataract surgery) eyes.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Difference in pro- inflammatory cytokine levels between patients undergoing a pIOL explantation in combination with a cataract surgery compared to patients only undergoing cataract surgery in aqueous humour. | up to 12 months after surgery
  Cytokines of interest are IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, TNF-α, MMP9. Detection will be in pg/mL.

SECONDARY OUTCOMES:
Correlation between inflammatory biomarkers (cytokines) in the aqueous humour and in tears | up to 12 months after surgery
  The following assay will be used: MSD multiplex pro-inflamatory kit.
Progress of EC loss after combined IF-pIOL explantation and cataract surgery compared to cataract surgery as a single procedure. | up to 12 months after surgery
  Progress will be measured with non-contact specular microscopy which will be the same for all patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No